CLINICAL TRIAL: NCT00108316
Title: SERT Affinity Determinants in Antidepressant Outcomes
Brief Title: Determinants in Antidepressant Outcomes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study PI resigned
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: MHBS-003-02S
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2013-09-27 (Estimated); Status verified 2013-09

CONDITIONS: Depression
Keywords: Depressive Disorder; DNA; Serotonin
MeSH Terms: conditions — Depression; Depressive Disorder | interventions — Fluoxetine

ARMS (1):
- Arm 1 (Other)
  Interventions: Drug: Fluoxetine (Liquid Prozac)

INTERVENTIONS:
Drug: Fluoxetine (Liquid Prozac)

SUMMARY:
This study is designed to understand if a biological measurement, of how platelets respond to serotonin (a chemical in the blood sometimes referred to as SERT), can provide information that will determine an "ideal dose," one specifically tailored for each individual's chemistry. The biological measurement will be obtained by testing a blood sample. There will be approximately 120 control subjects expected for enrollment.

DETAILED DESCRIPTION:
OBJECTIVE: The objective of this dose-ranging three-arm study of fluoxetine is to study the kinetics of the serotonin transporter in platelets and relate this to antidepressant response by comparing the manipulation of serotonin and platelet measure to standard treatment as it now exists.

RESEARCH PLAN: The project will examine two methods of dose adjustment of selective serotonin reuptake inhibitor (SSRI) treatment: The first method emulates the current standard clinical practice, i.e., titrating the dosage based upon the subject's current depression symptomatology (standard treatment arm). The second method utilizes the measurement of the Km to create a dosage tailored to the individual to approach the optimum treatment Kapp (biological treatment arm). Additionally, the placebo arm will control for treatment failure and high placebo response. This application is a double-blind, placebo controlled, randomized, dose ranging study in male and female outpatients with Major Depressive Disorder. The proposed study will take place over a period of 12 weeks recruiting 117 subjects (in order to achieve 90 completers, 30 in each arm, assuming 30% dropout rate) over a five year period who are diagnosed with Major Depression according to DSM-IV criteria. Following a 1 week screening period during which safety assessments are completed and evaluated and the Km and dosage are calculated, the subjects will be blindly randomized in a 1:1:1 ratio to either the standard treatment, the biological arm or the placebo arm. Subjects will return to the clinic at weeks 4, 8, and 12 for ratings and platelet Km determinations. Response will be measured and dosage adjustment will be made at weeks 4 and 8. A final determination of response will be made at week 12.

METHODS: Responders will be identified according to conventional criteria will be defined as those subject who 1) have a 50% or more improvement from baseline scores, as measured on the Hamilton Depression Scale (HAM-D), 2) no longer meet Major Depressive criteria according to DSM-IV; and 3) score < 10 on the HAM-D 17 item or <15 on the 24-item HAM-D. The efficacy measures will be the Hamilton Depression Scale (HAM-D): The seventeen item scale is designed to measure depression level; Montgomery-Asberg Depression Rating Scale (MADRS): A scale designed to provide additional subjective information to determine depressive symptoms; The Profile of Mood States (POMS) and the Cloninger Temperament Character Index (TCI) are patient rated scales which measure feelings and personality traits. The safety parameters include physical examinations, vital signs, collection of adverse events, and 12-lead electrocardiogram (ECG) and clinical laboratory assessments.

CLINICAL RELEVANCE: Previous studies have indicated fluoxetine is an effective treatment for depression. This study is designed to provide additional information concerning the methods for determining dose. Potentially, the information gained from this research may provide a more cost-effective way of finding an effective dose than the trial and error approach generally used.

ELIGIBILITY:
Inclusion Criteria:

* A current episode satisfying DSM-IV criteria for Major Depressive Disorder (except controls).
* No psychotropic medication during the previous 2 weeks before baseline (no SSRIs or SNRIs for previous 3 months).
* A current depression score of 20 or greater on the 24-item Hamilton Depression Scale (patients).
* Willingness and ability to give informed consent.
* Age 18 and up.

Exclusion Criteria:

* Cardiovascular disease; subjects w/ myocardial infarcts within the past 3 months, heart failure, or other evidence of compromised cardiac function
* Uncontrolled hypertension: systolic blood pressure > 160, or diastolic > 95
* Previously noted thyroid disease, unless clinically euthyroid for 2 or more months.
* Endocrine disease or exogenous hormones except HRT for postmenopausal women.
* Women not using an effective method of birth control (barrier method, oral contraceptives and/or IUD), pregnant or lactating women.
* Women with menometrorrhagia, premenstrual dysphoric disorder (PMDD), or premenopausal hysterectomized women with intact ovaries, or without HRT.
* Subjects who require concomitant psychotropic medications. Psychotropic medication during the previous 2 weeks before baseline, 3 months for SSRIs or SNRIs, or 4 months for depot neuroleptics.
* Evidence of clinically significant gastrointestinal, hepatic, renal, endocrine, ophthalmologic, neurologic, cardiovascular or hematological disease including anemia, hemophilia, or significant liver disease.
* History of intolerable side effects to the proposed treatment.
* Patients who have ever met DSM-IV criteria for any psychosis, schizophrenia, bipolar disorder, organic brain syndrome or any other primary Axis I major psychiatric disorder other than major depression. Controls must be without past history of depression.
* Patients who meet DSM-IV criteria for any substance abuse during the past 2 months or dependence during the last 6 months, including positive urine drug screens.
* History of priapism
* Subjects who are starting a new psychotherapy program during the 16 weeks of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2004-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Rausch, MD, Principal Investigator — VA Medical Center, Augusta
Locations (1):
- VA Medical Center, Augusta, Augusta, Georgia, United States